CLINICAL TRIAL: NCT00355537
Title: A Randomised, Double Blind, Placebo-controlled Parallel Study to Test the Effect of Testosterone Treatment on Peripheral Vascular Disease in Hypogonadal Men With Type 2 Diabetes Mellitus
Brief Title: Testosterone Replacement in Diabetes With Vascular Disease (Version 2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barnsley Hospital (Other)
Responsible Party: Prof Hugh Jones, Barnsley Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BDGH 237
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus; Peripheral Vascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Vascular Diseases | interventions — Testosterone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator)
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Testosterone — Sustanon- intramuscular testosterone 200mg every 2 weeks
  Arms: Active
Drug: 0.9% saline — Saline injection intramuscular every 2 weeks
  Arms: Placebo

SUMMARY:
Diabetes is a major cause of peripheral vascular disease(PVD) and is associated with male hypogonadism. Diabetes and PVD are both associated with arterial stiffness and intima -media thickness which are also related to severity of the clinical syndrome of PVD. Artificially induced hypogonadism results in increasing arterial stiffness whilst testosterone is known to improve risk factors for vascular disease and act as a vasodilator. The purpose of this pilot study is to assess the effect of testosterone treatment on PVD arterial stiffness and intima-media thickness in men with type 2 diabetes and hypogonadism,

ELIGIBILITY:
Inclusion Criteria:

* Male patients greater than 18 years of age
* Type 2 Diabetes Mellitus
* Serum testosterone less than 11 nmol/L on two consecutive samples taken on different days
* Peripheral vascular disease as defined by ABPI less than 0.92 and ischaemic leg pain (claudication or rest pain) or distal complications (non-healing arterial foot ulcer or gangrene
* Agreement to maintain antihypertensive and anti-lipid treatments at prior doses during 3 months of study
* Ability to give written informed consent after verbal and written explanation in the English Language
* Ability to comply with all study requirements

Exclusion Criteria:

* Current or previous breast cancer
* Current or previous prostate cancer
* Raised prostate specific antigen or abnormal per rectal examination unless prostate cancer excluded after specialist urology opinion
* Severe symptoms of benign prostatic hypertrophy ('prostatism')
* Treatment with testosterone in the 3 months prior to the trial
* Investigational drug treatment in the 3 months prior to the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The effect of testosterone replacement on arterial stiffness measured by ultrasound derived index B of the femoral artery in men with a combination of DM, PVD and hypogonadism. | 3 months

SECONDARY OUTCOMES:
The effect of testosterone on intima-media thickness of the femoral artery measured by ultrasound . | 3 months
The effect of testosterone on peripheral circulation in legs affected by PVD as measured by transcutaneous oxygen saturation in the feet of the study population. | 3 months
The effect of testosterone on PVD as measured by ankle-brachial-pressure-indices (ABPI) . | 3 months
The effect of testosterone on markers of vascular risk; blood pressure, serum-lipid levels, weight, waist circumference, body fat percentage, urinary micro-albumin concentration and C reactive protein levels. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Jones, Principal Investigator — Barnsley Hospital NHS Foundation Trust
Locations (1):
- Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire, United Kingdom